CLINICAL TRIAL: NCT05700994
Title: Peer Engagement in Methamphetamine Harm-Reduction With Contingency Management (PEER-CM)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Comagine Health (Other); Oregon Health Authority (Other)
Responsible Party: Principal Investigator, P. Todd Korthuis, MD, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: PEER-CM
Record Dates: First submitted 2023-01-17; First posted 2023-01-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Methamphetamine Abuse
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a cluster-randomized pragmatic trial using a hybrid type 1 effectiveness-implementation framework and stepped-wedge design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEER-CM (Experimental): Peer-facilitated contingency management (PEER-CM).
  Interventions: Behavioral: Peer Contingency Management
- Standard of Care (Active Comparator): Standard of care contingency management.
  Interventions: Behavioral: Standard of Care Contingency Management

INTERVENTIONS:
Behavioral: Peer Contingency Management — Participants allocated to peer-facilitated contingency management will receive incentives for achieving self-identified harm reduction goals set with peer specialists using a participant-driven harm reduction goal-setting process (e.g. completing overdose prevention and supply training, daily life goals, treatment and care goals, relationship and social support goals)
  Other Names: PEER-CM
  Arms: PEER-CM
Behavioral: Standard of Care Contingency Management — Participants allocated to standard of care contingency management will receive incentives for peer encounters.
  Other Names: Standard of Care
  Arms: Standard of Care

SUMMARY:
The main goal of this study is to tests the effect of incentivizing achievement of self-identified, personal harm reduction goals (Contingency management or CM) compared with standard of care (peer harm reduction service with incentives for peer visits) to increase the reach and effectiveness of methamphetamine (MA) harm reduction services.

DETAILED DESCRIPTION:
Using a hybrid type 1 effectiveness-implementation framework and stepped-wedge design, this study will randomize eighteen community-based peer harm reduction sites to provide contingency management incentives for achieving self-identified harm reduction goals set with peer specialists using a participant-driven harm reduction goal-setting process (e.g. completing overdose prevention and supply training, daily life goals, treatment and care goals, relationship and social support goals) versus standard of care contingency management (i.e. incentives for peer encounter attendance).

ELIGIBILITY:
Inclusion Criteria:

This intervention is at the site level. Community-based organization sites are eligible if they:

* Use peer support specialists to provide direct outreach and harm reduction services to people who use drugs
* Are willing to be trained in the two strategies for peer-facilitated contingency management

Clients who:

* Age 18 and older
* Any stimulant (methamphetamine, cocaine) use in the past 30 days
* Willing to accept peer services
* Willing to complete initial and follow-up assessments with peer
* Able to communicate in English or Spanish

Exclusion Criteria:

Community-based organization sites who:

* Do not use peer support specialists to provide direct outreach and harm reduction services to people who use drugs
* Are not willing to be trained in the two strategies for peer-facilitated contingency management

Clients who:

• Present any danger or threat of violence to peers

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1283 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants who overdose | 6 months from baseline
  Test the impact of incentives for achieving self-identified, personal harm reduction goals on the likelihood of overdose among people using methamphetamine at 6 months from enrollment identified through completed assessment.
Number of participants who achieve self-identified goals | 6 months from baseline
  Determine whether incentives for achieving self-identified, personal harm reduction goals increases engagement with harm reduction services at 6 months from enrollment identified through completed assessment.
Number of participants who engage in substance use disorder treatment | 6 months from baseline
  Determine whether incentives for achieving self-identified, personal harm reduction goals increases engagement with treatment services at 6 months from enrollment identified through completed assessment.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Comagine Health, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cooke A, Stack E, Peng L, Cook R, Hartzler B, Leichtling G, Hildebran C, Leahy JM, Payne KS, Kunkel LE, Hoffman K, Korthuis PT. The peers expanding engagement in stimulant harm reduction with contingency management study: a protocol paper. Addict Sci Clin Pract. 2025 Jun 10;20(1):48. doi: 10.1186/s13722-025-00577-8. PMID 40495203
- [Derived] Peng L, Stack E, Cooke A, Hartzler B, Cook R, Leichtling G, Hildebran C, Leahy J, Payne KS, Kunkel L, Hoffman K, Korthuis PT. Centering peers in design and training for a peer-delivered contingency management program for self-identified harm reduction and treatment goals. Harm Reduct J. 2025 May 6;22(Suppl 1):72. doi: 10.1186/s12954-025-01213-z. PMID 40329274